CLINICAL TRIAL: NCT06422637
Title: INFORM: A Prospective Interventional Study on Early Screening for Lung Cancer Using Liquid Biopsy
Brief Title: A Prospective Interventional Study on Early Screening for Lung Cancer Using Liquid Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ES-2024-025-02
Record Dates: First submitted 2024-05-14; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Liquid Biopsy for Early Screening of Lung Cancer
Keywords: Lung Cancer; Liquid Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): By collecting 2,972 peripheral blood samples from a natural population baseline, a comprehensive analysis of the fragmentomic characteristics of cfDNA was conducted based on whole-genome sequencing (WGS) of plasma cfDNA.
  Interventions: Diagnostic Test: Liquid Biopsy Early Screening
- control group (No Intervention): 2972 individuals were enrolled from the general population for routine LDCT screening.

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy Early Screening — An early screening model for lung cancer aids in identifying individuals with early-stage lung cancer. Those with positive indications of lung cancer will subsequently undergo confirmatory clinical assessments using Low-Dose Computed Tomography (LDCT) in sequence. Ultimately, a definitive diagnosis of lung cancer is established through surgical and pathological examination.
  Arms: Intervention group

SUMMARY:
This project aims to establish the MERCURY pilot screening program as part of the "Love Lung Project," employing a novel concept of lung cancer screening with the assistance of low-dose computer tomography (LDCT). By using clinical pathology as the gold standard, it will parallelly compare the performance (with a sensitivity of ≥90%) of the MERCURY early lung cancer screening model against the LDCT-only screening group within the "Love Lung Project." Ultimately, the objective is to reduce the proportion of overtreatment, achieve earlier staging, and extend patient survival, thus enhancing clinical value.

DETAILED DESCRIPTION:
This study is the first international prospective interventional study for lung cancer screening. It designates the "Love Lung Program" using Low-Dose Computed Tomography (LDCT) screening as the control group and the MERCURY screening group as the intervention group. Participants from the general population were enrolled and randomly assigned to either group in a 1:1 ratio. The MERCURY group plans to collect baseline peripheral blood samples from 2,972 individuals for whole genome sequencing (WGS) based on plasma circulating free DNA (cfDNA). This will facilitate a comprehensive analysis of the fragmentomics characteristics of cfDNA. Through the MERCURY early lung cancer screening model, individuals potentially at early stages of lung cancer will be identified. Those showing positive signs will subsequently undergo sequential LDCT to further confirm lung cancer status, eventually confirmed via surgery or pathology. To minimize ethical risks, the negative cases will receive additional LDCT after three months to further confirm their lung status. The control group under the "Love Lung Program" will follow standard LDCT screening procedures with the same number of participants; those with positive LDCT results will undergo clinical diagnosis, while those with negative results will only be followed up for lung status. Relying on the "Love Lung Program," the objective is to establish a new concept of lung cancer screening that precedes with MERCURY screening assisted by LDCT diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 40 years old and less than 75 years old, regardless of gender.
* Sign the informed consent form.

Exclusion Criteria:

* Pregnant women;
* Individuals currently diagnosed with any tumors other than lung cancer, or who have a history of cancer;
* Those who have undergone LDCT/CT screening within the past 1-3 years;
* Individuals currently suffering from a febrile illness, or who have had an acute inflammatory disease episode requiring internal medicine treatment within the last 14 days prior to blood draw;
* Individuals who have taken corticosteroids orally or through intravenous injection within the 14 days prior to blood draw;
* Organ transplant recipients or those who have previously received a non-autologous (allogeneic) bone marrow or stem cell transplant;
* Individuals in poor health or not suitable for blood drawing;
* Any other clinically significant disease or condition considered by the researchers to potentially affect adherence to the protocol, impact the patient's ability to provide informed consent, or render the patient unsuitable for participation in the clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5944 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value | 2 years
  When a test result indicates that a patient is positive, the probability that the true condition is positive.

SECONDARY OUTCOMES:
Detection rate of non-stage 0 lung cancer within 2 years | 2 years
  the proportion of patients diagnosed with lung cancer through clinical pathology in both the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — Department of Medical Oncology of Respiratory, Guangxi Medical University Cancer Hospital
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
publish an article